CLINICAL TRIAL: NCT01414283
Title: A Phase 1 Dose-escalation Study of PSMA ADC in Subjects With Progressive, Castration-resistant, Metastatic Prostate Cancer
Brief Title: Prostate-specific Membrane Antigen Antibody-Drug Conjugate in Subjects With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSMA ADC 1301
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PSMA ADC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: PSMA ADC

INTERVENTIONS:
Drug: PSMA ADC — PSMA ADC administered IV

SUMMARY:
Prostate-specific Membrane Antigen Antibody-Drug Conjugate (PSMA ADC) 1301 is an open-label, dose-escalation phase 1 study of PSMA ADC administered IV in subjects with progressive, castration-resistant, metastatic prostate cancer that has progressed after prior taxane therapy. For all subjects, PSMA ADC will be administered in four repeating cycles.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of progressive, castration-resistant, metastatic prostate cancer.
2. Prior chemotherapy regimens, one of which contains taxane.
3. Eastern Cooperative Oncology Group status of 0 or 1

Exclusion Criteria:

1. Clinically significant cardiac disease or severe debilitation pulmonary disease
2. Evidence of an active infection requiring ongoing antibiotic therapy
3. Any prior treatment with any other therapy targeting PSMA
4. History of drug and/or alcohol abuse

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-10; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of PSMA ADC | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Israel, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States